CLINICAL TRIAL: NCT05493891
Title: Testing the Association Between Low Back Pain Intensity and Core Muscle Strength in Women Who Underwent Cesarean or Vaginal Deliveries
Brief Title: Low Back Pain Intensity and Core Muscle Strength After Different Delivery Modes
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Lecturer of Physical Therapy for Women's Health, South Valley University
Other Study IDs: Core muscle strength
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain and Core Muscle
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: 18 participants have been exposed to cesarean delivery
  Interventions: Other: Visual analogue scale (VAS); Device: Pressure Biofeedback Unit (PBU)
- Group B: 18 participants have been exposed to vaginal delivery
  Interventions: Other: Visual analogue scale (VAS); Device: Pressure Biofeedback Unit (PBU)

INTERVENTIONS:
Other: Visual analogue scale (VAS) — VAS is a reliable and valid method for assessing the intensity of low back pain (LBP)
Device: Pressure Biofeedback Unit (PBU) — PBU is a valid and reliable instrument for measuring the maximal voluntary isometric contraction of both lumbar multifidus and transversus abdominis muscles (core muscle strength)

SUMMARY:
Cesarean delivery (CD) may trigger an increase in low back pain (LBP) intensity and induce core muscle weakness. This study will assess the correlation between low back pain intensity and core muscle strength of transverse abdominis and Lumbar multifidus among women who underwent CD and compare it with those who experienced vaginal delivery.

DETAILED DESCRIPTION:
Cesarean delivery (CD) is one of the most common surgical procedures in obstetrics, and it is also one of the oldest medical procedures. The rise in the rate of cesarean sections is one of the most striking hallmarks of modern obstetrics.

In Egypt, the prevalence of CD has increased dramatically over the last decade, with the most recent Egypt Demographic and Health Survey (EDHS) reporting a rate of 52 percent, implying that cesarean sections may be overused or utilized for improper reasons.

The two deep local core muscles are the transversus abdominis and the lumbar multifidus muscles. The definition of Core muscle strength is the active ability of these muscles to not only produce but also, maintain stresses to provide stability for the spine through management of the intra-abdominal pressure.

LBP prevalence in mothers undergoing cesarean delivery was higher compared to its counterpart in mothers undergoing vaginal delivery. The related mechanisms for LBP during the postpartum period following cesarean or vaginal deliveries may be overweight and obesity, postural adaptations, and stressful positions that mothers assume during either delivery or lactation.

ELIGIBILITY:
Inclusion Criteria:

1. All women are either primiparous or multiparous.
2. Their ages ranged from 18 to 35 years.
3. All participants had a body mass index (BMI) of not more than 29.5, and a waist-to-hip ratio of not more than 1.
4. Participants were assessed between the 6th week to the 12th week postnatal.
5. All participants were able to continue all assessment procedures.
6. They were medically stable.

Exclusion Criteria:

1. Women who were below 18 years old or above 35 years old.
2. Women who had a (BMI) above 29.5 or a waist-to-hip ratio above 1.
3. Women who did not continue all assessment procedures.
4. Women who had a past history of specific LBP as those who were diagnosed with spondylolisthesis, lumbar disc prolapse, or structural scoliosis.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Because this study is specific to women's health physical therapy specialty
Study Population: 36 participants participated in our study, and were classified into 2 groups; (group A) represents 18 mothers undergoing cesarean birth, and (group B) represents 18 mothers undergoing normal vaginal birth.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2023-08-05 (Actual)

PRIMARY OUTCOMES:
The intensity of LBP | Assessment will be done 6-12 weeks after Cesarean OR Vaginal deliveries
  The intensity of low back pain is a standardized method to quantify the severity of low back pain
The maximal voluntary isometric contraction of the transversus abdominis muscle | Assessment will be done 6-12 weeks after Cesarean or Vaginal Deliveries
  The maximum voluntary isometric contraction (MVIC) is an objective standardized method with high reliability used to evaluate and quantify muscle strength
The maximal voluntary isometric contraction of the lumbar multifidus muscle | Assessment will be done 6-12 weeks after Cesarean or Vaginal Deliveries
  The maximum voluntary isometric contraction (MVIC) is an objective standardized method with high reliability used to evaluate and quantify muscle strength
The correlation coefficient between low back pain intensity and core muscle strength | Assessment will be done 6-12 weeks after Cesarean or Vaginal Deliveries
  The correlation coefficient between two variables of outcome is a valid statistical method to the association between them

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barber EL, Lundsberg LS, Belanger K, Pettker CM, Funai EF, Illuzzi JL. Indications contributing to the increasing cesarean delivery rate. Obstet Gynecol. 2011 Jul;118(1):29-38. doi: 10.1097/AOG.0b013e31821e5f65. PMID 21646928
- [Background] Abdel-Tawab N, Oraby D, Hassanein N, and El-Nakib S. Cesarean Section Deliveries in EGYPT: Trends, Practices, Perceptions and Cost, Cairo: Population Council. 2018.
- [Background] Mhyre JM, Sultan P. General Anesthesia for Cesarean Delivery: Occasionally Essential but Best Avoided. Anesthesiology. 2019 Jun;130(6):864-866. doi: 10.1097/ALN.0000000000002708. No abstract available. PMID 30985305
- [Background] Ring L, Landau R, Delgado C. The Current Role of General Anesthesia for Cesarean Delivery. Curr Anesthesiol Rep. 2021;11(1):18-27. doi: 10.1007/s40140-021-00437-6. Epub 2021 Feb 24. PMID 33642943
- [Background] Traynor AJ, Aragon M, Ghosh D, Choi RS, Dingmann C, Vu Tran Z, Bucklin BA. Obstetric Anesthesia Workforce Survey: A 30-Year Update. Anesth Analg. 2016 Jun;122(6):1939-46. doi: 10.1213/ANE.0000000000001204. PMID 27088993
- [Background] Malatova R, Rokytova J, Stumbauer J. The use of muscle dynamometer for correction of muscle imbalances in the area of deep stabilising spine system. Proc Inst Mech Eng H. 2013 Aug;227(8):896-903. doi: 10.1177/0954411913486078. Epub 2013 May 1. PMID 23636767
- [Background] Faries MD, Greenwood M. Core training: stabilizing the confusion. Strength and conditioning journal. 2007 Apr 1;29(2):10.
- [Background] Parikh S, Suchi J. Prevalence of low back pain and its impact on quality of life in post-partum women. International Journal of Scientific Research. 2016; 7:14342-8.
- [Background] MacArthur C, Lewis M, Knox EG, Crawford JS. Epidural anaesthesia and long term backache after childbirth. BMJ. 1990 Jul 7;301(6742):9-12. doi: 10.1136/bmj.301.6742.9. PMID 2143425